CLINICAL TRIAL: NCT05464498
Title: Evaluation of Collagen-based Medical Device Treatment Combined With Physiotherapy in Subjects With Achilles Tendinopathy. Multicenter Randomized Clinical Investigation; AKITENMED STUDY.
Brief Title: Evaluation of Collagen-based Medical Device Treatment Combined With Physiotherapy in Subjects With Achilles Tendinopathy.
Acronym: AKITENMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guna S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDG20180000
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-11

CONDITIONS: Tendinopathy; Insertional Achilles Tendinopathy; Achilles Tendinopathy; Peritendinitis
Keywords: Eccentric strengthening; Collagene Medical Device; Physiotherapy; Peritendinous area; Infiltration; Type I collagen; Eccentric strengthening protocol; Pain Visual Analog Scale; 12-Item Short Form Survey; Victorian Institute of Sport Assessment- Achilles questionnaire
MeSH Terms: conditions — Tendinopathy; Tenosynovitis; Osteogenesis Imperfecta, Type IV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MD-Tissue Medical Device (Experimental): Group A which, alongside physiotherapy (eccentric strengthening protocol) will receive MD-Tissue Collagen Medical Device.
  Interventions: Device: MD-Tissue Collagen Medical Device; Other: eccentric strengthening protocol
- Eccentric strengthening protocol (Other): Group B who will only perform physiotherapy (eccentric strengthening protocol).
  Interventions: Other: eccentric strengthening protocol

INTERVENTIONS:
Device: MD-Tissue Collagen Medical Device — MD-Tissue (GUNA, Milan-Italy) Composition per 2 ml: collagen 100 micrograms Excipients: Ascorbic acid, Magnesium gluconate, Pyridoxine hydrochloride, Riboflavin, Thiamine hydrochloride, NaCl, Water for injection.
  Subjects will be treated with No. 6 peri-tendon injections (2 infiltrations per week for three weeks).
  Arms: MD-Tissue Medical Device
Other: eccentric strengthening protocol — Group B which, will implement only physiotherapy (eccentric strengthening protocol)

SUMMARY:
Achilles tendinopathy is a condition characterized by inflammation of the Achilles tendon. Achilles tendinopathies are classified into insertional tendinitis and noninsertional tendinitis. Insertional tendinitis involves the lower part of the tendon, where the tendon inserts at the level of the calcaneus, and can affect even patients who are not particularly athletically active. Noninsertional tendinitis occurs when the fibers in the middle portion of the tendon are affected, affects young and athletic people the most, and has a high incidence (30-50%) in middle-aged individuals.

Considering that there are no strong evidence-based guidelines in the area of treatment of achilles tendinopathy, the aim of this research project is to understand through a multicenter, randomized clinical investigation the impact of treatment with a porcine collagen-based medical device administered in the peri-tendon area in combination with physiotherapy on pain reduction and functional improvement of the investigated tendon.

DETAILED DESCRIPTION:
In view of the morpho-structural changes that characterize Achilles tendinopathy, the use of injectable medical devices such as Collagen Medical Devices might find therapeutic indication. For some years now, in fact, the use of injectable medical devices based on porcine collagen and ancillary substances of natural origin (Collagen Medical Devices GUNA) has been introduced in the treatment of painful and degenerative pathologies of the locomotor system, which allow a more effective and specific placement of collagen in situ with the function of vehiculation and stabilization.

The purpose of this research project is to understand through a multicenter, randomized clinical study investigation the impact of treatment with a porcine Collagen-based Medical Device called MD-Tissue, administered in the peri-tendon area, in combination with physiotherapy on pain reduction and functional improvement of the investigated tendon.

The multicenter, randomized clinical investigation is prospective, and will have a total duration of 8 weeks.

After enrollment, subjects will be randomized and assigned to two experimental groups:

* Group A which, alongside physiotherapy (eccentric strengthening protocol) will receive MD-Tissue Collagen Medical Device.
* Group B which, will implement only physiotherapy (eccentric strengthening protocol).

Variables will be assessed at baseline (T0 time), after 1 week (T1), after 2 weeks (T2), after 3 weeks (T3), at the end of the injection treatment, and 6 weeks after enrollment (T6/FU). A further evaluation will be carried out after 2 weeks and after 8 weeks T8/FU from the start of the investigation study.

After enrollment, subjects in both groups will begin a physiotherapy course (eccentric strengthening protocol), lasting 6 weeks. Each session will consist of stretching exercises of the Achilles tendon.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 70 years;
* Subjects with tendon pain for not more than 24 weeks;
* Subjects with clinically diagnosed and ultrasonographically confirmed insertional/noninsertional/mystic tendinopathy;
* Subjects with a VISA A score between 50 and 75;
* VAS ≥ 5;
* Subjects able to understand and answer the SF12 questionnaire;
* Subjects able to understand and sign the informed consent.

Exclusion Criteria:

* subjects who have had surgery in the investigated area or lower extremity;
* subjects who have previously undergone physiotherapy.
* subjects with autoimmune diseases;
* subjects with peripheral neuropathy;
* subjects with calcific tendinopathy
* subjects with pain of direct traumatic origin;
* subjects with local/systemic infections;
* subjects with neoplastic diseases;
* subjects with gout;
* subjects on corticosteroid treatment at the time of enrollment;
* subjects who have used corticosteroids or fluoroquinolones in the three months prior to enrollment;
* subjects who have used NSAIDs in the week prior to enrollment;
* subjects who are pregnant and lactating;
* subjects with contraindications to acetaminophen use;
* allergy to porcine collagen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
Assessment of the VISA-A questionnaire score at week 8, ranging from 0 to 100 points, where 100 points represents a healthy tendon. | Weeks 8
  The primary end point will be assessed at week 8 and will involve: Assessment of the VISA-A questionnaire score at time weeks 8 compared to day 0. A difference between the two groups of 12 out of 100 points on the questionnaire can be considered clinically significant.
  We measured the VISA-A score (ranging from 0 to 100 points, where 100 points represents a healthy tendon.

SECONDARY OUTCOMES:
Assessment of the VISA-A (Victorian Institute of Sport Assessment- Achilles) questionnaire score at T3 and T6 weeks, ranging from 0 to 100 points, where 100 points represents a healthy tendon. | Weeks 3, weeks 6.
  Evaluation of VISA-A score at time weeks 3 and weeks 6 compared to day 0. We measured the VISA-A score (ranging from 0 to 100 points, where 100 points represents a healthy tendon
Assessment of the VAS (Visual Analogue Scale) at time weeks 3, weeks 6 and weeks 8, allows the patient to define pain intensity along a line from 0 to 10 cm (100 mm). | Weeks 3, weeks 6, weeks 8
  Assessment of the VAS (Visual Analogue Scale) at time weeks 3, weeks 6 and weeks 8 compared to day 0.
  Visual Analogue Scale (VAS) allows the patient to define pain intensity along a line from 0 to 10 cm (100 mm). One end indicates no pain 'no pain' while the other represents maximum pain 'maximum pain'.
Evaluation of the SF12 (Item Short Form Survey) questionnaire at times weeks 3, weeks 6 and weeks 8 determinated the phisical condition and mental healthy functioning. | Weeks 3, weeks 6 and weeks 8.
  Evaluation of the SF12 (Item Short Form Survey) questionnaire at time weeks 3, weeks 6 and weeks 8 compared to day 0.
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning A score of 50 or less o has been recommended as a cut-off to determine a physical condition; while a score of 42 or less may be indicative of 'clinical depression.
  The questionnaire needs to be supported by a statistical programme for further analysis.
Evaluation of the fraction of subjects in each group achieving Minimal Clinical Disease (MCD) considering that the MCD of the VISA-A questionnaire is 18.5 (90% MCD). | Day 0, week 1, weeks 2,weeks 3, weeks 6 and weeks 8.
  Evaluation of the fraction of subjects in each group achieving Minimal Clinical Disease (MCD) considering that the MCD of the VISA-A questionnaire is 18.5 (90% MCD), after treatment and study duration.
Assessment of analgesic drug unit consumption based on clinical diary | Weeks 3,weeks 6 and weeks 8.
  Assessment of analgesic drug unit consumption based on clinical diary at time weeks 3, weeks 6 and weeks 8, (paracetamol 1000 mg. will be used as "rescue dose" in case of onset/recurrence of pain).
Evaluation of the fraction of subjects in each group who drop out early in relation to Adverse Events (AE/SAE/SUSAR) | Day 0, week 1,weeks 2,weeks 3,weeks 6 and weeks 8.
  Evaluation of the fraction of subjects in each group who drop out early in relation to Adverse Events (AE/SAE/SUSAR

CONTACTS AND LOCATIONS:
Overall Officials: Paoloni PM Marco, Prof, Principal Investigator — U.O.C. Medicina Fisica e Riabilitativa dell'AOU "Policlinico Umberto I°" Piazzale Aldo Moro, 5 00185 Roma
Locations (1):
- U.O.C. Medicina Fisica e Riabilitativa dell'AOU "Policlinico Umberto I°", Roma, RO, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT05464498/Prot_001.pdf